CLINICAL TRIAL: NCT01859325
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled Study of a Multi-Antigen DNA Vaccine Prime Delivered by In Vivo Electroporation, rVSV Booster Vaccine in HIV-Infected Patients Who Began Antiretroviral Therapy During Acute/Early Infection
Brief Title: Therapeutic Vaccine for HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Auro Vaccines LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 130141; 13-I-0141
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2018-05

CONDITIONS: HIV; Therapeutic Vaccine
Keywords: HIV-MAG pDNA Prime; HIV Therapy; Therapeutic Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): HIV-MAG pDNA vaccine prime will be administered at a dose of 3000 g (1500 g of the HIV-1 gag/pol plasmid and 1500 g of the HIV-1 net/tat/vif, env plasmid) at week 0, 4, 12, and 36. Each construct of HIV-MAG pDNA vaccine (1500 g each) will be mixed and combined with 1000 g of the IL-12 pDNA adjuvant. The resulting mixture will be divided into 2 IM injections and administered as 0.75 mL IM injection in the left deltoid and 0.75 mL IM injection in the right deltoid with EP using the TDS device. IL-12 pDNA adjuvant will be mixed with the HIV-MAG pDNA vaccine prime, as noted above, and administered at a dose of 1000 g (500 g in each IM injection) at week 0, 4, 12, and 36. rVSV HIV gag booster vaccine--The total dose, 1x107 pfu, will be administered as 1 mL (5x106 pfu) IM injection in the left deltoid and 1 mL (5x106 pfu) IM injection in the right deltoid at week 24 and 48.
  Interventions: Biological: rVSV; Biological: IL-12 pDNA adjuvant; Biological: HIV-Mag pDNA
- Placebo (Placebo Comparator): Placebo for the IL-12 pDNA adjuvant and HIV-MAG pDNA vaccine (sodium chloride for injection, USP 0.9%) will be administered as 0.75 mL IM injection in the left deltoid and 0.75 mL IM injection in the right deltoid at weeks 0, 4, 12, and 36 with EP using the TDS device. Placebo for the rVSV HIV gag (sodium chloride for injection, USP 0.9%) will be administered as 1 mL IM injection in the left deltoid and 1 mL IM injection in the right deltoid at week 24 and 48.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: rVSV — Attenuated recombinant vesicular stomatitis virus containing HIV-1 gag gene
  Arms: Vaccine
Biological: IL-12 pDNA adjuvant — plasmid DNA containing human IL-12 gene
  Arms: Vaccine
Biological: HIV-Mag pDNA — plasmid DNA vaccine containing genes encoding multiple HIV-1 proteins
  Arms: Vaccine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Background:

- In most people who have human immunodeficiency virus (HIV), the immune system cannot control or cure the infection. Antiretroviral therapy drugs can keep the amount of HIV virus low for a long time. However, this treatment does not remove the virus from the body. In the vast majority of patients antiretroviral therapy also will not protect the body from the virus once treatment stops. Researchers want to see if therapeutic vaccination can help people with HIV. Therapeutic vaccination means giving vaccines to treat an infection that someone already has (HIV, in this case). It may help the body's immune system attack the infection. This study will look at different measures of HIV infection after receiving either therapeutic vaccination or a placebo.

Objectives:

- To see whether therapeutic vaccination is safe and can affect how the body responds to HIV infection.

Eligibility:

- Individuals between 18 and 65 years of age who have HIV and are taking antiretroviral therapy drugs.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* During the screening visit and throughout the study until week 56, participants will continue to take their HIV medications.
* Participants will be divided into two groups. One group will have the study vaccines. The other will have a placebo.
* The first study vaccine or placebo will be given in weeks 4, 12, and 36. The second study vaccine or the placebo will be given in weeks 24 and 48. Blood samples and other tests will be given at each visit.
* After the study visit at week 56, participants will stop their HIV medications until week 72. From weeks 58 through 72, they will come in every 2 weeks for study visits; each visit will take about 1 hour to complete. These visits will look at the body s response to the vaccines and their HIV viral load. After week 72, participants will re-start their HIV medications.
* There will be follow-up study visits from weeks 76 to 96, with blood tests and other studies.

DETAILED DESCRIPTION:
The advent of combination antiretroviral therapy (cART) has dramatically improved the clinical outcome in human immunodeficiency virus (HIV)-infected individuals through sustained reduction in viral replication. However, it has become clear that cART alone cannot eradicate HIV in infected individuals, likely in part due to the persistence of viral reservoirs in peripheral blood and various tissue compartments. Consequently, a major thrust of HIV research over the past several years has been to develop therapeutic strategies that can eliminate persistent viral reservoirs and boost host immunity to control viral replication upon discontinuation of cART. Therapeutic HIV vaccination is one approach that could potentially achieve these goals through vaccine-induced improvement in HIV-specific immune responses and/or by direct reactivation of HIV-specific CD4+ memory T cells that harbor latent HIV. An effective therapeutic vaccine could augment immunologic control of HIV infection and potentially obviate the need for chronic cART.

The current study is an exploratory randomized, 2-arm (1:1), double-blind, placebo-controlled trial evaluating the safety and efficacy of an HIV-1 multiantigen plasmid DNA (HIV-MAG pDNA) vaccine prime in combination with an interleukin-12 plasmid DNA (IL-12 pDNA) adjuvant delivered by in vivo electroporation followed by a recombinant vesicular stomatitis virus vector containing the HIV-1 gag gene (rVSV HIV gag) booster vaccine in subjects on cART who started therapy during acute or early HIV infection.

Subjects will be randomized to receive placebo or the HIV-MAG pDNA (3000 g) vaccine prime and IL-12 pDNA adjuvant (1000 g) at week 0, 4, 12, and 36, and the rVSV HIV gag booster vaccine (1x107 plaque-forming units) at week 24 and 48. The HIV-MAG pDNA vaccine prime and IL-12 pDNA adjuvant will be administered as 2 IM injections, 1 into each deltoid, with electroporation using the Ichor TDS device, while the rVSV HIV gag booster vaccine will be administered as 2 conventional IM injections, 1 into each deltoid. After the week 56 visit, all subjects will undergo an analytical treatment interruption to determine if the vaccination strategy results in an improved immune control of viral replication, as evidenced by a blunted or absent rebound in HIV plasma viremia. All subjects will be followed through week 96 for safety and efficacy parameters.

The study population includes HIV-infected adults who began cART during acute or early infection. Subjects must be receiving an effective cART regimen, with a CD4 cell count of >450 cells/mm3 at screening, and they must have documented viral suppression below the limit of detection for greater than1 year. The rationale for testing the study vaccine regimen in this subject population is because these individuals may have a relatively preserved immune function, which could be augmented by therapeutic vaccination.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age, 18-65 years.
  2. Institution of cART within 12 weeks of being diagnosed with acute or early HIV-1 infection.

     Acute HIV-1 infection is defined as:
     1. Detectable plasma HIV-1 RNA levels of greater than 2000 copies/mL with a negative result from an HIV-1 EIA, or
     2. Positive result from an HIV-1 EIA with a negative or indeterminate result from an HIV-1 western blot that subsequently evolves to a confirmed positive result, or
     3. Negative result from an HIV-1 EIA within the past 4 months and HIV-1 RNA levels of greater than 400,000 copies/mL, in the setting of a potential exposure to HIV-1.

     Early HIV-1 Infection is defined as:
     1. Negative result from an HIV-1 EIA within 6 months prior to a positive result from an HIV-1 EIA and an HIV-1 western blot.
     2. Negative result from a rapid HIV-1 test within 1 month prior to a positive result from an HIV-1 EIA and an HIV-1 western blot.
     3. Presence of low level of HIV antibodies as determined by having a positive EIA or a positive Western blot with a non-reactive detuned EIA according to a serologic testing algorithm for recent infection.
  3. CD4+ cell count greater than 450 cells/mm3 at screening.
  4. Documentation of continuous cART treatment with suppression of plasma viral level below the limit of detection for greater than 1 year. Subjects with a single blip (i.e., detectable viral levels on cART) prior to randomization may be included provided they satisfy the following criteria:

     1. The blips are less than 400 copies/mL, and
     2. Succeeding viral levels return to levels below the limit of detection on subsequent testing.
  5. Willingness to undergo ATI.
  6. Laboratory values within pre-defined limits at screening:

     * Absolute neutrophil count greater than 1,000/mm3.
     * Hemoglobin levels greater than 10.0 g/dL for men and greater than 9.0 g/dL for women.
     * Platelet count greater than 100,000/mm3.
     * Prothrombin time (PT) and partial thromboplastin time (PTT) less than 1.5 upper limit of normal (ULN).
     * Estimated or a measured creatinine clearance rate of greater than 60 mL/min as determined by the NIH Clinical Center laboratory.
     * AST and ALT levels of less than 2.5 x ULN.
  7. Willingness to have samples stored for future research.
  8. Women of childbearing potential must have a negative pregnancy test result.

     * They must agree to use an adequate form of contraception:

       * Hormonal contraception.
       * Male or female condoms with or without a spermicidal
       * Diaphragm or cervical cap with a spermicidal.
       * Intrauterine device.

EXCLUSION CRITERIA:

1. Allergy to amide-type local anesthetics (bupivacaine (Marcaine), lidocaine (Xylocaine), Mepivacaine (Polocaine/Carbocaine), etidocaine (Duranest), prilocaine (Citanest, EMLA cream).
2. Chronic hepatitis B, as evidenced by a positive test for hepatitis B surface antigen (HBsAg), or chronic hepatitis C virus (HCV) infection, as evidenced by a positive test for HCV RNA. Subjects with a positive test for HCV antibody and a negative test for HCV RNA are eligible.
3. Changes in cART regimen due to virologic breakthrough.
4. HIV immunotherapy or vaccine(s) received within 1 year prior to screening.
5. Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) received within 4 weeks prior to study entry.
6. Interruption of cART for greater than 3 months since its initiation. 8. Any active malignancy that may require systemic chemotherapy or radiation therapy.
7. Pregnancy or planned pregnancy during the study period or breastfeeding.
8. Any active malignancy that may require systemic chemotherapy or radiationtherapy.
9. Immunosuppressive medications received within 6 months before the first study vaccination (Not excluded: (1) corticosteroid nasal spray for allergic rhinitis; (2) topical corticosteroids for mild, uncomplicated dermatitis; or (3) oral/parenteral corticosteroids administered for non-chronic conditions not expected to recur (length of therapy less than or equal to10 days, with completion in greater than or equal to 30 days prior to enrollment).
10. Evidence of hepatic decompensation in subjects with cirrhosis: history of ascites, hepatic encephalopathy, or bleeding esophageal varices, or screening laboratory results with any of the following:

    1. International normalized ratio of greater than or equal to1.5 x ULN.
    2. Serum albumin less than 3.2 g/dL.
    3. Serum total bilirubin greater than 1.8 x ULN, unless history of Gilbert's disease or deemed related to treatment with atazanavir.
11. History or other clinical evidence of:

    1. Significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction, significant arrhythmia).
    2. Severe illness, malignancy, immunodeficiency other than HIV, or any other conditions that, in the opinion of the investigator, would make the subject unsuitable for the study.
    3. AIDS-defining condition.
12. Known allergy or sensitivity to the components of the investigational therapy.
13. History of significant cardiac arrhythmia (e.g., supraventricular tachycardia, ventricular tachycardia, and atrial fibrillation/flutter).
14. Active drug or alcohol use or any dependence other pattern of behaivor that, in the opinion of the investigator, would interfere with adherence to study requirements.
15. Any active systemic inflammatory or autoimmune disease or condition.
16. Presence of implanted electronic medical device (e.g., pacemaker, implantable cardiac defibrillator) or surgical/traumatic metal implant in the upper limb and/or upper torso.
17. Neurological or neuropsychiatric disorder that may interfere with the assessment of safety (e.g., frequent recurring headaches, for example, a pattern of greater than 1 headache/month affecting activities of daily living/work, frequent or severe/complicated migraines, cluster headaches); or history of encephalitis, narcolepsy, stroke with sequelae, moderate/severe major depressive disorder, moderate/severe bipolar disorder, seizure disorder.
18. Deltoid skinfold measurements (by caliper) of greater than 40 mm.
19. Body mass index greater than 40.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2017-02-26 (Actual); Study Completion 2017-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volberding PA, Deeks SG. Antiretroviral therapy and management of HIV infection. Lancet. 2010 Jul 3;376(9734):49-62. doi: 10.1016/S0140-6736(10)60676-9. PMID 20609987
- [Background] Richman DD, Margolis DM, Delaney M, Greene WC, Hazuda D, Pomerantz RJ. The challenge of finding a cure for HIV infection. Science. 2009 Mar 6;323(5919):1304-7. doi: 10.1126/science.1165706. PMID 19265012
- [Background] Trono D, Van Lint C, Rouzioux C, Verdin E, Barre-Sinoussi F, Chun TW, Chomont N. HIV persistence and the prospect of long-term drug-free remissions for HIV-infected individuals. Science. 2010 Jul 9;329(5988):174-80. doi: 10.1126/science.1191047. PMID 20616270
- [Result] Sneller MC, Justement JS, Gittens KR, Petrone ME, Clarridge KE, Proschan MA, Kwan R, Shi V, Blazkova J, Refsland EW, Morris DE, Cohen KW, McElrath MJ, Xu R, Egan MA, Eldridge JH, Benko E, Kovacs C, Moir S, Chun TW, Fauci AS. A randomized controlled safety/efficacy trial of therapeutic vaccination in HIV-infected individuals who initiated antiretroviral therapy early in infection. Sci Transl Med. 2017 Dec 6;9(419):eaan8848. doi: 10.1126/scitranslmed.aan8848. PMID 29212716
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-I-0141.html

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-Mag/IL-12 & rVSV Vaccine: HIV-MAG pDNA vaccine prime will be administered at a dose of 3000 g (1500 g of the HIV-1 gag/pol plasmid and 1500 g of the HIV-1 net/tat/vif, env plasmid) at week 0, 4, 12, and 36. Each construct of HIV-MAG pDNA vaccine (1500 g each) will be mixed and combined with 1000 g of the IL-12 pDNA adjuvant. The resulting mixture will be divided into 2 IM injections and administered as 0.75 mL IM injection in the left deltoid and 0.75 mL IM injection in the right deltoid with EP using the TDS device. IL-12 pDNA adjuvant will be mixed with the HIV-MAG pDNA vaccine prime, as noted above, and administered at a dose of 1000 g (500 g in each IM injection) at week 0, 4, 12, and 36. rVSV HIV gag booster vaccine--The total dose, 1x107 pfu, will be administered as 1 mL (5x106 pfu) IM injection in the left deltoid and 1 mL (5x106 pfu) IM injection in the right deltoid at week 24 and 48.
- Excluded: Participants not meeting inclusion criteria or declined to participate.
Period: Overall Study
Arm/Group | HIV-Mag/IL-12 & rVSV Vaccine | Placebo | Excluded
Started | 15 | 16 | 2
Completed | 12 | 12 | 2
Not Completed | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-Mag/IL-12 & rVSV Vaccine | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 11 | 18
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Related Adverse Events in Subjects Who Began cART During Acute or Early HIV-1 Infection.
Description: The rate of occurrence of grade 3 or higher AEs, including serious adverse events (SAEs) that per standard criteria (see safety section) are:
  At least possibly related to the test article, and Definitely NOT related to a factor other than the test article This is to evaluate safety and tolerability of the study vaccines.
Time Frame: 48 weeks
Population: All subjects who received vaccine or placebo
Measure: Number; unit: Related Adverse Events
Arm/Group | HIV-Mag/IL-12 & rVSV Vaccine | Placebo
Number analyzed (Participants) | 14 | 15
Related Adverse Events | 0 | 0

2. Secondary Outcome: HIV-1 Viral Load Following Antiretroviral Treatment Interruption (ATI).
Description: The difference in HIV-1 viral load at the end of the ATI between the vaccine and placebo groups. Levels of plasma viremia in the vaccine and placebo groups were compared using the Wilcoxon rank sum test at the end of treatment interruption periods to determine the antiviral efficacy of the therapeutic vaccine regimen. The limit of detection of plasma viremia was 40 copies/ml of HIV RNA.
Time Frame: 72 weeks
Population: All subjects who received vaccine or placebo
Measure: Median (Inter-Quartile Range); unit: copies/ml
Arm/Group | HIV-Mag/IL-12 & rVSV Vaccine | Placebo
Number analyzed (Participants) | 14 | 15
copies/ml | 4932 [513 to 22577] | 3170 [467 to 7025]
Statistical Analysis 1: Comparison: HIV-Mag/IL-12 & rVSV Vaccine vs Placebo; Samples size based on published data on populations of early treated patients undergoing ART interruption. The power based on a 2-sample t-test with a 2-tailed alpha of .05 and a total sample size of 30 is approximately 91% to detect a 1.25 log10 reduction in the rebound plasma viremia between vaccine and placebo groups; Test type: Superiority; p = 0.406, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -.36, 95% CI 2-sided [-1.41 to 0.67]

ADVERSE EVENTS:
Time Frame: 96 weeks
Arm/Group | HIV-Mag/IL-12 & rVSV Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/16
Other Adverse Events (participants affected / at risk) | 15/15 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-Mag/IL-12 & rVSV Vaccine (N=15) | Placebo (N=16)
Cellulitis (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-Mag/IL-12 & rVSV Vaccine (N=15) | Placebo (N=16)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 2
Oral disorder (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 5 | 2
Fatigue (General disorders) | 11 | 7
Injection site erythema (General disorders) | 2 | 5
Injection site pain (General disorders) | 15 | 15
Injection site swelling (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gonorrhoea (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tinea versicolour (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 5
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Injury (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 2
Blood bicarbonate abnormal (Investigations) | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 3
C-reactive protein increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 7
Headache (Nervous system disorders) | 6 | 5
Migraine (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Toe amputation (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT01859325/Prot_SAP_000.pdf
  • Informed Consent Form (2015-08-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT01859325/ICF_001.pdf